CLINICAL TRIAL: NCT03582059
Title: A Prospective, Double Blind, Cross Over, Pilot Study to Evaluate EEG Changes in Patients' Undergoing Spinal Cord Stimulation(SCS) With High Frequency and Burst Frequency for Failed Back Surgery Syndrome(FBSS).
Brief Title: Electroencephalographic Changes in Spinal Cord Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PM16/84656
Record Dates: First submitted 2016-09-23; First posted 2018-07-10 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Single blind, randomized cross over study at a single centre
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group meeting inclusion criteria group 1 (Other): Patients meeting the inclusion criteria in the first 10 days of entering trial and are randomised to first intervention.
  Interventions: Procedure: High Frequency Spinal cord stimulation; Procedure: Burst Frequency Spinal cord stimulation
- Patient group meeting inclusion criteria group 2 (Other): Patient group meeting inclusion criteria after 10 days and are allocated second intervention.
  Interventions: Procedure: High Frequency Spinal cord stimulation; Procedure: Burst Frequency Spinal cord stimulation

INTERVENTIONS:
Procedure: High Frequency Spinal cord stimulation — An electrode will be implanted into the patients back. A defined stimulation patter will be applied. The patient will be randomised to received 7-10 days of high frequency stimulation.
Procedure: Burst Frequency Spinal cord stimulation — An electrode will be implanted into the patients back. A defined stimulation patter will be applied. The patient will be randomised to received 7-10 days of burst frequency stimulation.

SUMMARY:
Spinal cord stimulation by means of an electrode in the back is used to treat patients with persistent chronic pain after back surgery. Based on the stimulation patterns, there are mainly three different technologies available - conventional, burst frequency and the high frequency. It is known that the traditional frequency works through the lateral system of pain pathways in the spinal cord to cause pain reduction. Electroencephalographic(tracing of brain activity) recording of patients using burst have shown an additional effect on an adjacent medial pain pathway which decreases the attention to pain. We want to therefore find out if high frequency stimulation also has an effect on the same pathways. 20 patients who have persistent neuropathic chronic pain after previous spinal surgery, would be eligible to have this treatment as part of their normal care. They will be randomly chosen to undergo a 2 week cycle of high frequency and 2 weeks of burst stimulation. We will record EEG's, pain scores and scores measuring attention to pain and compare findings. All patients will be recruited at the Leeds Pain and Neuromodulaton centre and the EEg analysis will be done by a research team based in Belgium. We hope that the study will improve our understanding of how different stimuation waveforms used for spinal cord stimulation work. We hope to have recruited all 20 patients in a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

* I. Patient is 18 years of age or older and has given written informed consent. II. Has persistent chronic predominant low back pain of neuropathic origin, with or with out radiculopathy, for a minimum of 6 months as per NICE Tag 0159. III. Patient has had previous spinal surgery at least > 6 months ago. IV. Numerical rating scale Scale (NRS) back pain score of at least 5 at baseline V. Confirmation of pain from neuropathic origin as per NICE guidance TAG 0159 VI. Total daily dose of opioids equivalent to ≤120mg of Morphine VII. In the investigators opinion the patient is a suitable candidate for SCS. VIII. Patient is willing to comply with the requirements of the study

Exclusion Criteria:

* I. Patient has mechanical spine instability based on flexion/extension testing of lumbar spine (documented in the last 6 months) II. Patient is pregnant, or pregnancy is suspected or planned within the first six months of the study timeframe.

III. Patient has a cardiac pacemaker, automatic defibrillator, or any other implanted device, which will make the trial impossible. IV. Allergy to device components or drugs to be used in the intended procedure. V. Medical co-morbidities that preclude surgical intervention. VI. Patient is incapable of understanding or responding to the study questionnaires VII. Patient is incapable of understanding or operating the patient programmer handset.

VIII. Patient is morbidly obese (BMI ≥ 40). IX. Patient is simultaneously participating in another device or drug study within the last 30 days.

X. Patient is on more than 120 mg of morphine a day. XI. Patient has a spinal fracture, tumour or infection. XII. Clinical evidence of cauda equina syndrome. XIII. Progressive neurologic deficit. XIV. Patient has epilepsy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Electrencephalographic patterns generated | 60 mins
  Pain measured according to pain vigilance and awareness questionnaire (PVAQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No